CLINICAL TRIAL: NCT05094414
Title: Urology Department, Hualien Tzu Chi Hospital, Hualien, Taiwan
Brief Title: Using Oral Valacyclovir to Treat Patients With Refractory IC/BPS
Acronym: VARIC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government); Hualien Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Hann-Chorng Kuo, Urology department, Hualien Tzu Chi General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOST 109 2314 B 303 024
Record Dates: First submitted 2021-10-14; First posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Pain, Chronic; Urge Incontinence; Overactive Bladder Syndrome; Quality of Life
MeSH Terms: conditions — Chronic Pain; Urinary Incontinence, Urge | interventions — Valacyclovir

STUDY DESIGN:
Intervention Model Description: The IC/BPS patients would be investigated for baseline clinical symptoms questionnaire including VAS, QoL, ICPI, ICSI, and OSS. All of our patients would receive open-label oral valacyclovir 500 mg twice per day for 4 weeks. We estimate to enroll 30 IC/BPS patients. The overall improvement of current therapy would be assessed with Global Response Assessment (GRA).The GRA, VAS, and any adverse effect would be investigated in the telephone interview. After the full 4 weeks treatment, the patients would be asked to back to our clinic. All symptoms questionnaire (GRA, VAS, QoL, ICPI, ICSI, and OSS) and adverse effect would be evaluated again. The patients would be asked to provide urine sample again. The primary endpoint of this study is the GRA at 4 weeks. The secondary endpoints include the changes of VAS, VAS, QoL, ICPI, ICSI, and OSS between baseline and end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Valacyclovir — oral valacyclovir 500 mg twice per day for 4 weeks

SUMMARY:
Interstitial cystitis/bladder pain syndrome (IC/BPS) is a collective term referring to disorders which is characterized by lower urinary tract symptoms, including bladder pain/discomfort, frequent urination without evidence of bacterial infection. The etiology of IC/BPS is still uncertain, and most current treatment for IC/BPS are only symptoms control. Our previous study revealed Epstein-Barr virus (EBV) infection presented in the IC/BPS bladders and involved the pathogenesis. Hence, using anti-viral medication valacyclovir for the patients with IC/BPS might have clinical efficacy.

DETAILED DESCRIPTION:
We would like to conduct a prospective study to evaluate to therapeutic effect of oral valacyclovir for the patients with IC/BPS. The diagnosis of IC/BPS was made through following the clinical symptom index of the American Urological Association guideline. The IC/BPS patients with concurrent urological diseases, such as neurogenic voiding dysfunction, ketamine cystitis or acute bacterial cystitis in recent one month would be excluded. The IC/BPS patients with possibility of pregnancy also would be rule out.

At first, the enrolled patients would be investigated for urinary analysis and culture to rule out current bacteriuria. The enrolled patients would receive a comprehensive medical history review. A pregnancy test would be performed for women of childbearing potential. The patients would be asked to provide urine sample to urinary virus investigation before the treatment. The IC/BPS patients would be investigated for baseline clinical symptoms questionnaire including VAS, QoL, ICPI, ICSI, and OSS. The parameters in the VUDS report also would be record. The Informed consent would be obtained from all individual participants before the intervention. Due to higher bioavailability, we would use valacyclovir in this study. The dose of valacyclovir we use is according to previous valacyclovir study for genital HSV infection. [18] According previous valacyclovir study for chronic recurrence herpesvirus infection disease, long-term therapy of oral valacyclovir < 1000mg/day should be effective and safe; the safety profiles of valacyclovir and placebo were similar. All of our patients would receive open-label oral valacyclovir 500 mg twice per day for 4 weeks.

We estimate to enroll 30 IC/BPS patients with evidence of EBV infection in bladder into this study. After the beginning of valacyclovir therapy, the patients would receive a telephone interview to evaluated current symptoms changes at first and second weeks. The overall improvement of current therapy would be assessed with Global Response Assessment (GRA) (3: symptoms free, 2: >50% symptoms improvement, 1: 25-50% symptoms improvement, 0: 0-25% symptoms improvement, -1: symptoms worse). The GRA, VAS, and any adverse effect would be investigated in the telephone interview. After the full 4 weeks treatment, the patients would be asked to back to our clinic. All symptoms questionnaire (GRA, VAS, QoL, ICPI, ICSI, and OSS) and adverse effect would be evaluated again. The patients would be asked to provide urine sample again. The primary endpoint of this study is the GRA at 4 weeks. The secondary endpoints include the changes of VAS, VAS, QoL, ICPI, ICSI, and OSS between baseline and end of the study. The following figure showed the study flow diagram.

ELIGIBILITY:
Inclusion Criteria:

* patients with IC/BPS

Exclusion Criteria:

* patients with neurogenic bladder
* patients with bladder outlet obstruction
* patients with lymphoma
* patients with bacteria cystitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Global Response Assessment (GRA) | 1 month
  3: symptoms free, 2: >50% symptoms improvement, 1: 25-50% symptoms improvement, 0: 0-25% symptoms improvement, -1: symptoms worse

SECONDARY OUTCOMES:
VAS | 1 month
  VAS scale for pain
OSS | 1 month
  O'Leary-Sant Symptom Index

CONTACTS AND LOCATIONS:
Locations (1):
- Hualien Tzu Chi Hospital, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kuo HC, Peng CW, Jiang YH, Jhang JF. Urinary Viral Spectrum in Patients with Interstitial Cystitis/Bladder Pain Syndrome and the Clinical Efficacy of Valacyclovir Treatment. Biomedicines. 2024 Feb 26;12(3):522. doi: 10.3390/biomedicines12030522. PMID 38540138